CLINICAL TRIAL: NCT06072443
Title: AURORA Study-A Transformative Approach Utilizing Behavioral Economics, Education, and Data Science to Support Patients Initiating PrEP With Retention-in-care and Medication Persistence
Brief Title: AURORA Study-A Transformative Approach to Support PrEP Medication Persistence
Status: Recruiting | Type: Observational
Sponsor: WV Health Right, Inc. (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 220084
Record Dates: First submitted 2023-09-01; First posted 2023-10-10 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
Keywords: PrEP; HIV Prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAB-LA PrEP Cohort: Prescribed CAB-LA PrEP as standard of care or current user of CAB-LA PrEP
  Interventions: Behavioral: Digital Health Companion (mobile App)
- Oral PrEP Cohort: Prescribed oral PrEP as standard of care or current user of oral PrEP
  Interventions: Behavioral: Digital Health Companion (mobile App)

INTERVENTIONS:
Behavioral: Digital Health Companion (mobile App) — Participants will complete education modules, health literacy evaluations, and PRO assessments in the Digital Health Companion.

SUMMARY:
This study is designed to test the hypothesis that, compared to oral PrEP, use of CAB-LA in underserved populations in a real-world setting supported by a digital health companion program will be associated with greater medication adherence, persistence, retention-in-care, and improved PROs. Patients in the study will receive current standard care for HIV prevention and be offered enrollment in the digital health companion program.

Goal of the study is to evaluate medication adherence and persistence in patients receiving CAB-LA vs oral PrEP and who engage with a digital health companion program.

DETAILED DESCRIPTION:
The study will evaluate the extent to which real-world use of CAB-LA for PrEP in underserved populations impacts PrEP adherence, persistence, retention-in-care, and PROs compared with oral PrEP. Additionally, the study will examine the implementation of a digital health companion program that leverages education and behavioral economics to support patients on PrEP, and assess clinician perspectives as well as barriers to, and facilitators for implementation of CAB-LA in a patient-centered medical home.

Primary Objective To evaluate medication adherence and persistence in patients receiving CAB-LA vs oral PrEP and who engage with a digital health companion program

Secondary Objectives Evaluate retention-in-care in patients receiving CAB-LA vs oral PrEP Evaluate PROs (including PrEP Medication Satisfaction, PrEP Acceptance, P Evaluate the acceptability, appropriateness, and helpfulness of a digital health companion program for PrEP Evaluate the acceptability, barriers to, and facilitators for implementation of CAB-LA

Study Design The research project follows a hybrid effectiveness-implementation research design, with the primary aim focused on evaluation of PrEP adherence, persistence and retention-in-care with CAB-LA compared with oral PrEP, and secondary aims focused on evaluating patient-reported outcomes (PROs), implementation of a digital health intervention to support adherence and persistence, and evaluating contextual factors around implementation of CAB-LA. The proposed study will utilize a digital health intervention with behavioral health economics and patient education from PRIME and Reciprocity to evaluate the adoption and implementation of a Digital Health Companion for PrEP adherence and persistence. The implementation aims of the study will leverage the RE-AIM framework as follows: Assessment of the digital health intervention will focus primarily on individual-level dimensions of RE-AIM, including reach and effectiveness. For example, in assessing reach of the digital health intervention, participant demographics will be compared to the intended audience to evaluate the extent to which populations with high unmet needs were engaged. Conversely, assessment of the implementation of CAB-LA will focus on system-level dimensions of RE-AIM, such as qualitative assessments of barriers to and facilitators for implementation of CAB-LA. In addition, evaluation of PROs will be informed by a review of validated instruments, including HIVSTQ (HIV Treatment Satisfaction Questionnaire), SMSQ (Study Medication Satisfaction Questionnaire), I-TAQ (Injection Treatment Acceptance Questionnaire), ACCEPT (Chronic Treatment Acceptance Questionnaire), and the PrEP Stigma Scale, with survey items tailored to evaluate PrEP acceptance, satisfaction, and perceptions of PrEP-related stigma for both the CAB-LA and oral PrEP arms.

Description of Study Procedures Before any screening procedure is performed, informed consent will be obtained. Labs will be taken at baseline and months 3, 5, 7, 9, and 11 for the CAB-LA cohort and at baseline and months 3, 6, 9, and 12 for the Oral PrEP cohort. Participants will complete a baseline evaluation and be introduced to a support group at baseline. Patients will complete assessments within the Reciprocity App. Clinicians will complete assessments outside of the app. Patients in both cohorts will complete baseline demographic surveys in month 0, patient reported outcomes (PRO) data collection set 1 in months 1, 5, and 11 and PRO data collection set 2 in months 3, 9, and 12. Patients in the CAB-LA PrEP cohort will complete persistence assessments in months 1, 3, 5, 7, 9, and 11. Patients in the Oral PrEP cohort will complete persistence assessments every month from months 1 through 12. Clinic staff will complete surveys at baseline, month 6, month 12, and at the end of the study.

Medication Persistence Definition: Continue to take medicines over time independent of adherence to the PrEP medication regimen.

Persistence Assessment CAB-LA The proportion of participants who received at least one PrEP injection who remained on injectable PrEP or oral bridging at months 3 and 11 measured by the self-report assessment and validated with claims data.

Persistence Assessment Oral PrEP The proportion of participants who initiated oral PrEP who remained on oral PrEP at months 3 and 12 measured by the self-report assessment and validated with claims data. period.

Adherence Definition: Taking PrEP in line with medical advice/using PrEP appropriately (critical for efficacy) .

Adherence Assessment CAB-LA

Adherence to the dosing schedule will be assessed at month 3 (early adherence) and end of study by:

A) Estimating the number of individuals who missed one or more consecutive injections without taking daily oral bridging PrEP while not on CAB-LA injections and mean and median number of injections missed during a 6- and a 12-month period.

B) Estimating the number of individuals who received the injections seven or more days later than their scheduled injection visit and the mean and median duration of delayed injections.Adherence Assessment Oral PrEP

Adherence to the dosing schedule will be assessed at months 3 (early adherence) and 12 by:

A) Estimating the number of individuals who reported three or more days of oral PrEP missed and the mean and median number of days they missed.

B) Estimating the number of individuals who had a gap of >90 days between the end of the days of supply of a dispensing and the start date of the next fill.

Patient Reported Outcomes Patient Reported Outcomes Set 1: PrEP Medication Satisfaction, PrEP-Related Stigma, Acceptability of Intervention Measure (AIM) Patient Reported Outcomes Set 2: PrEP Acceptance, Intervention Appropriateness Measure (IAM) Helpfulness of the education modules and Health Literacy Evaluation

Clinician Instruments Baseline Provider Survey Information About You and Your Patients Acceptability of Intervention Measure (AIM) Intervention Appropriateness Measure (IAM) Feasibility of Intervention Measure (FIM) Barriers and Facilitators for Implementation of Long-Acting

Cabotegravir for PrEP Follow-up Provider Survey Information About You and Your Patients Acceptability of Intervention Measure (AIM) Intervention Appropriateness Measure (IAM) Feasibility of Intervention Measure (FIM) Barriers and Facilitators for Implementation of Long-Acting Cabotegravir for PrEP

Standard of Care Visits The standard of care for patient visits will not be affected. The patients will only be given additional surveys to complete.

Follow-Up Visits CAB-LA PrEP cohort: 2nd PrEP injection at month 1; follow-up labs and PrEP injections in months 3, 5, 7, 9, and 11.

Oral PrEP cohort: follow-up labs and prescription refills in months 3, 6, 9, and 12.

Switching between PrEP regimens .To be included in final data analysis, participants cannot switch between PrEP regimens before 6-months duration of initial PrEP.

PrEP Discontinuation Participants will be deemed as having discontinued PrEP if they miss more than 3 consecutive months for PrEP.

Participants will be called, texted and emailed for three consecutive months before considered them as discontinued.

STI Screening and Management Participants will receive STI screening at baseline and at every follow up clinic visit. Participants will be screened if they present with any type of symptoms that warrant STI testing. If a participant tests positive for an STI other than HIV, they will receive guideline-directed therapy at the discretion of their

HCP at WVHR. Suspected or Confirmed HIV Infection HIV screening will occur a minimum as recommended for every 2 months with CAB-LA (same time as injections) and every 3 months for oral PrEP.

PrEP Choice Counselling Patients will be counseled on the benefits and risks of both oral PrEP and PrEP injections. The selection of PrEP option will be done as the standard of care through shared-decision with the patient.

Possible Participant Pathways There will only be two observational cohort arms. Patients will either be placed into the injectable PrEP arm or the oral PrEP arm based on their baseline prescription.

Adherence Strategies Patients on oral PrEP will be encouraged to set a daily reminder on their smart phone as an alarm at the time their dose is due.

Patients on injectable PrEP will set a monthly calendar reminder on the day/time their injection is due.

Retention Strategies Follow-up appointments will be set up and conveyed at each appointment. Reminder calls will be made by a staff member a few days before the appointment.

Interventions: PrEP Initiation and Digital Health Companion Program Participants will be enrolled in the CAB-LA and Oral PrEP cohorts. Participants in the CAB-LA cohort will receive their first dose of the PrEP injection at month 0. Injections will also be administered in months 1, 3, 5, 7, 9, and 11. Participants in the Oral PrEP cohort will have their prescription filled at month 0, 3, 6, 9, and 12. The schedule of dosing is presented in Figure 6a.

Participants in both cohorts will complete education modules and health literacy evaluations in the Reciprocity App in months 2, 4, 6, 8, and 10 as presented in Figure 6a. Education Modules include PrEP Medicines (month 2), Protecting Yourself from HIV, STIs, and other infections (month 4), Building a Support System for HIV Prevention Month 6: Being an Active Participant in Your Own Care (month 8), and Overcoming Stigma and Becoming a Health Advocate (month 10).

Adherence to oral PrEP and reasons for PrEP discontinuation will be assessed through brief behavioral surveys every month after the initiation of PrEP. Barriers to adherence to CAB-LA injections and reasons for PrEP discontinuation will be assessed through brief behavioral surveys at months 1, 3, 5, 7, 9, and 11.

Implementation Outcomes for the Mobile App Acceptability of the mobile app to support patients in taking PrEP will be measured by the Acceptability of Intervention Measure (AIM) at months 1, 5, and 11. Appropriateness of the mobile app to support patients in taking PrEP will be measured by the Intervention Appropriateness Measure (IAM) at months 3, 9, and 12.

Clinic Staff Acceptability, Appropriateness, and Feasibility of Providing Long-acting Cabotegravir Injections Acceptability of the process for providing long-acting cabotegravir injections will be assessed by the Acceptability of Intervention Measure (AIM). Appropriateness of the process for providing long-acting cabotegravir injections will be assessed by the Intervention Appropriateness Measure (IAM).

Feasibility of long-term use of cabotegravir injections will be assessed by the Feasibility of Intervention Measure (FIM). Willingness to sustain provision of long-acting cabotegravir injections and barriers to and facilitators for provision of long-acting cabotegravir injections will be assessed through a brief survey. The clinic staff surveys will be administered at baseline, month 6, month 12, and end of study.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of or current user of PrEP with CAB-LA, daily FTC/TDF, or daily FTC/TAF prescribed in accordance with the WVHR standard of care practices (based practices on CDC PrEP 2021 Clinical Practice Guidelines) by a licensed HCP
* PrEP dispensed by WVHR pharmacy
* Access to a smart phone

Exclusion Criteria:

* Receiving HIV PrEP care outside of WVHR
* Positive HIV diagnosis
* Contraindication to oral or injectable PrEP therapy
* Receiving oral bridging therapy prior to injectable PrEP therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving HIV prevention care at WVHR.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: Medication Adherence | 12-months
  Medication adherence will be calculated as the percentage of patients adherent to PrEP at months 3 and at the end of the study. The adherence percentages will be assessed by using WV Pharmacy dispensement data for the CAB-LA and Oral PrEP cohorts. Adherence will be assessed by calculating the medication possession ratio for Oral PrEP to quantify the number of oral PrEP doses missed and the percentage of participants who missed one or more injections or received injections outside the 7 day window for the target date of their CAB-LA injection. The final calculation will represent the percentage of patients in each cohort who were adherent to all prescribed PrEP doses.

SECONDARY OUTCOMES:
EFFICACY: Retention in Care | 12-months
  Retention in care will be calculated in patients receiving CAB-LA vs oral PrEP as the percentage of patients with an electronic medical record documented clinic visit within 30 days of their scheduled visit at months 3, 9 and 12 for the Oral PrEP cohort and at months 3, 9, and 11 for the CAB-LA cohort. The final calculation will represent the percentage of patients in each cohort who completed all scheduled clinic visits.
SATISFACTION: Patient Experiences with PrEP | 12-months
  Patient experiences with PrEP medications will be assessed through a questionnaire with patients selecting from a 5-point scale ranging "very dissatisfied" to "very satisfied" in 6 question domains. Percentages of patient reported satisfaction will be compared between Oral PrEP and CAB-LA cohorts.
QUALITY OF LIFE: Patient Experiences with PrEP-related stigma | 12-months
  Patient experiences with PrEP-related stigma will be assessed through a questionnaire with patients selecting from a 5-point scale ranging "completely disagree" to "completely agree" in 11 question domains. Percentages of patient reported agreement will be compared between Oral PrEP and CAB-LA cohorts.
SATISFACTION: Patient Experiences with mobile App | 12-months
  Patient experiences with mobile App will be assessed through a questionnaire with patients selecting from a 5-point scale ranging "5=completely disagree" to "1= completely agree" in 4 question domains. Percentages of patient reported agreement will be compared between Oral PrEP and CAB-LA cohorts.
ACCEPTABILITY: Provider Acceptability of Intervention Measure (AIM) | 12-months
  Provider experiences with mobile App intervention will be assessed through a questionnaire with providers selecting from a 5-point scale ranging "5=completely disagree" to "1= completely agree" in 4 question domains. Percentages of provider reported agreement will be calculated into percentages for each answer choice.
ACCEPTABILITY: Provider Intervention Appropriateness Measure (IAM) | 12-months
  Provider experiences with CAB-LA care will be assessed through a questionnaire with providers selecting from a 5-point scale ranging "5=completely disagree" to "1= completely agree" in 4 question domains. Percentages of provider reported agreement will be calculated into percentages for each answer choice.
FEASIBILITY: Provider Feasibility of Intervention Measure (FIM) | 12-months
  Provider experiences with feasibility of CAB-LA care will be assessed through a questionnaire with providers selecting from a 5-point scale ranging "5=completely disagree" to "1= completely agree" in 4 question domains. Percentages of provider reported agreement will be calculated into percentages for each answer choice.

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia Health Right, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YA, Tao G, Smith DK, Hoover KW. Persistence With Human Immunodeficiency Virus Pre-exposure Prophylaxis in the United States, 2012-2017. Clin Infect Dis. 2021 Feb 1;72(3):379-385. doi: 10.1093/cid/ciaa037. PMID 33527117
- [Background] Keyes J, Crouse EC, DeJesus E, Rolle CP. Determinants of pre-exposure prophylaxis (PrEP) persistence in a high-risk population in Central Florida. J Investig Med. 2021 Feb;69(2):397-401. doi: 10.1136/jim-2020-001352. Epub 2020 Dec 1. PMID 33262130
- [Background] Spinelli MA, Scott HM, Vittinghoff E, Liu AY, Gonzalez R, Morehead-Gee A, Gandhi M, Buchbinder SP. Missed Visits Associated With Future Preexposure Prophylaxis (PrEP) Discontinuation Among PrEP Users in a Municipal Primary Care Health Network. Open Forum Infect Dis. 2019 Feb 26;6(4):ofz101. doi: 10.1093/ofid/ofz101. eCollection 2019 Apr. PMID 30949540
- [Background] Krakower D, Maloney KM, Powell VE, Levine K, Grasso C, Melbourne K, Marcus JL, Mayer KH. Patterns and clinical consequences of discontinuing HIV preexposure prophylaxis during primary care. J Int AIDS Soc. 2019 Feb;22(2):e25250. doi: 10.1002/jia2.25250. PMID 30768762
- [Background] Weitzman PF, Zhou Y, Kogelman L, Rodarte S, Vicente SR, Levkoff SE. mHealth for pre-exposure prophylaxis adherence by young adult men who have sex with men. Mhealth. 2021 Jul 20;7:44. doi: 10.21037/mhealth-20-51. eCollection 2021. PMID 34345621
- [Background] Garrison LE, Haberer JE. Pre-exposure Prophylaxis Uptake, Adherence, and Persistence: A Narrative Review of Interventions in the U.S. Am J Prev Med. 2021 Nov;61(5 Suppl 1):S73-S86. doi: 10.1016/j.amepre.2021.04.036. PMID 34686294
- [Background] Woodcock A, Bradley C. Validation of the HIV treatment satisfaction questionnaire (HIVTSQ). Qual Life Res. 2001;10(6):517-31. doi: 10.1023/a:1013050904635. PMID 11789552
- [Background] Arnould B, Gilet H, Patrick DL, Acquadro C. Item Reduction, Scoring, and First Validation of the ACCEPTance by the Patients of their Treatment (ACCEPT(c)) Questionnaire. Patient. 2017 Feb;10(1):81-92. doi: 10.1007/s40271-016-0187-7. PMID 27456210
- [Background] Klein H, Washington TA. The Pre-Exposure Prophylaxis (PrEP) Stigma Scale: Preliminary findings from a pilot study. Int Public Health J. 2019;11(2):185-195. PMID 32089789
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT06072443/Prot_SAP_ICF_000.pdf